CLINICAL TRIAL: NCT00277329
Title: A Phase 2 Study of XL999 Administered Intravenously to Subjects With Non-Small-Cell Lung Cancer
Brief Title: Study of XL999 in Patients With Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to cardiac toxicities in the subejcts
Sponsor: Symphony Evolution, Inc. (Industry)
Responsible Party: Charles W. Finn, PhD, President and CEO, Symphony Evolution, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL999-204
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2010-02-22 (Estimated); Status verified 2010-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: XL999 — • The Study Treatment Period, in which subjects received a once-weekly, 4-hour intravenous (IV) infusion of XL999 at 2.4 mg/kg as outpatients for 8 weeks. Treatment was to be stopped at the occurrence of disease progression or unacceptable toxicity.

SUMMARY:
This clinical study is being conducted at multiple sites to determine the activity, safety, and tolerability of XL999 when given weekly to patients with non-small cell lung cancer (NSCLC). XL999 is a small molecule inhibitor of multiple kinases including VEGFR, PDGFR, FGFR, FLT-3, and Src, which are involved in tumor cell growth, formation of new blood vessels (angiogenesis), and metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with histologically confirmed NSCLC
* Prior treatment with a platinum- or taxane containing regimen
* Stage IIIB with malignant effusion, stage IV or recurrent NSCLC that is not amenable to curative therapy (either surgery or radiation therapy)
* Measurable disease according to Response Criteria for Solid Tumors (RECIST)
* ECOG performance status of 0 or 1
* Life expectancy ≥3 months
* Adequate organ and marrow function
* No other malignancies within 5 years
* Signed informed consent

Exclusion Criteria:

* Radiation to ≥25% of bone marrow within 30 days of XL999 treatment
* Use of any systemic anticancer therapy within 30 days of XL999 treatment
* More than 2 prior systemic cytotoxic chemotherapy regimens
* More than 1 prior agent targeted against VEGF or EGFR (eg, bevacizumab, erlotinib, or gefitinib)
* Subject has not recovered to ≤ grade 1 or to within 10% of baseline from adverse events due to other medications administered >30 days before study enrollment
* Uncontrolled and/or intercurrent illness
* History of or known brain metastases, current spinal cord compression, or carcinomatous meningitis
* Pregnant or breastfeeding females
* Known HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2005-12; Primary Completion 2007-08 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Response rate | Inclusion until disease progression
Safety and tolerability | Inclusion until 30 dyas post last treatment

SECONDARY OUTCOMES:
Progression-free survival | Inclusion until disease progression
Duration of response | Inclusion until disease progression
Overall survival | Inclusion until 180-Day Follow-up post last treatment or death
Pharmacokinetic (PK) and Pharmacodynamic (PD) parameters | Various time points during the 8-week Study Treatment Period in the second stage of the study

CONTACTS AND LOCATIONS:
Overall Officials: Paul Woodard, MD, Study Director — Exelixis
Locations (4):
- United States (4):
  - Hematology/Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Joliet Oncology-Hematology Associates, Ltd., Joliet, Illinois
  - Hematology-Oncology Associates of Rockland, Nyack, New York
  - Center for Oncology Research and Treatment, PA, Dallas, Texas